CLINICAL TRIAL: NCT06530225
Title: Are Louisiana Pharmacists PrEPared? Implementing Training and an Active PrEP (Pre-Exposure Prophylaxis) Prescribing Surveillance Program to Achieve Equity in Pharmacy Based PrEP Prescribing in Louisiana
Brief Title: Are Louisiana Pharmacists PrEPared? Implementing Training and an Active PrEP (Pre-Exposure Prophylaxis) Prescribing Surveillance Program
Status: Not yet recruiting | Type: Observational
Sponsor: Xavier University of Louisiana. (Other)
Collaborators: Louisiana Public Health Institute (Other)
Responsible Party: Sponsor
Other Study IDs: IRB1014-25
Record Dates: First submitted 2024-07-27; First posted 2024-07-31 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: HIV Prevention
Keywords: PrEP, HIV Prevention
MeSH Terms: interventions — Educational Status

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Community Based Pharmacies: Community based pharmacies throughout Louisiana will be enrolled in a cohort of trained pharmacies for PrEP prescriptions for patients seeking HIV prevention medication.
  Interventions: Other: Education and Mentoring for Prescribing Pharmacists

INTERVENTIONS:
Other: Education and Mentoring for Prescribing Pharmacists — Pharmacists enrolled in the PrEP prescribing cohort will receive implicit bias, health disparity and health equity training for HIV prevention. In addition, the pharmacists will receive mentorship and receive an implementation toolkit on best practices for PrEP prescribing.

SUMMARY:
Though broadening PrEP (Pre-Exposure Prophylaxis) availability to Louisiana pharmacies addresses key access issues for Louisiana's population, there is no current baseline data which explore current pharmacist and pharmacies' capacity to effectively provide PrEP therapy to patients who meet PrEP prescribing criteria. This study aims to explore1) Louisiana pharmacist and pharmacy capacity to provide PrEP under a state-based collaborative practice agreement, 2) a validated pharmacist education system addressing health disparities in PrEP prescribing and 3) the impact of state pharmacy based policies on equitable PrEP prescribing. Our central hypothesis is pharmacist trained in PrEP prescribing focusing on health disparities and implicit bias education and working with mentors in an implementation framework will have an increase in equitable PrEP prescribing

DETAILED DESCRIPTION:
The objective of this application is to create a statewide cohort of dispensing community-based pharmacists that are specifically trained to address health disparities in PrEP (Pre-Exposure Prophylaxis) prescribing. The specific aims of this application are:

Aim #1: Complete a rapid pharmacy landscape assessment on PrEP prescribing and maintenance from community pharmacies across Louisiana to measure frequency of PrEP seeking, prescribing and follow-up of PrEP initiation Hypothesis 1a: Pharmacists in rural parishes (counties) will have lower overall PrEP prescribing rates compared to their urban and suburban counterparts.

Hypothesis 1b: PrEP utilization patterns by African Americans, Hispanics and Women of all races will have a decreased lack of utilization PrEP compared to their white, male counterparts.

Aim #2: Measure the impact of a validated pharmacist PrEP training program on pharmacist competence and capacity in PrEP prescribing for CDC recognized target populations. The focus of the education will be addressing health disparities and implicit bias in PrEP prescribing.

Hypothesis 2:Pharmacists who complete the implicit bias and cultural competence training will report a 20% increase in baseline confidence and competence in PrEP prescribing for target vulnerable communities.

Aim #3: Measure the impact of an implementation science community-pharmacy based intervention on addressing PrEP prescribing among women, African-Americans and Hispanics. The impact of the program will implement a state-based PrEP surveillance program housed in the College of Pharmacy comparing PrEP prescribing patterns among trained pharmacists vs clinic based prescribing (control) as provided by the consortium of health network data housed at the Louisiana Public Health Institute.

Hypothesis 3a: Trained pharmacists will have a 15% increase in pharmacy PrEP dispensing from baseline vs non-trained pharmacists in the research network.

Hypothesis 3b: Pharmacy PrEP prescribing among trained pharmacists will represent a 20% increase in minority based prescribing, specifically African-American, compared to current health network clinic prescribing patterns.

ELIGIBILITY:
Inclusion Criteria:

* Community pharmacists in Louisiana providing PrEP prescriptions.

Exclusion Criteria:

* None

Ages: 24 Years to 99 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All practicing community pharmacists who are interested in a PrEP education course on equitable PrEP prescribing to address health disparities among the target patient population.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2026-05-01 (Estimated); Primary Completion 2029-04-30 (Estimated); Study Completion 2030-04-30 (Estimated)

PRIMARY OUTCOMES:
PrEP Prescribing | May 1, 2025- April 30, 2029
  Number of PrEP prescriptions dispensed from pharmacy (Scale PrEP prescription/1,000 total prescriptions in 30 day period)
Pharmacists' Knowledge and Confidence in PrEP prescribing | May 1, 2025- April 30, 2026
  Pharmacists will complete a pre and post-test on knowledge and confidence in PrEP prescribing to target populations. Knowledge will be scored on a graded scale of 0 (lowest to 100 (highest). Confidence will be scored on a Likert Scale (1 - least confident, 5 most confident)

CONTACTS AND LOCATIONS:
Locations (1):
- Xavier University of Louisiana, New Orleans, Louisiana, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified, conglomerate data will be provided upon request.
Supporting Information: Study Protocol, SAP
Time Frame: 5/1/25 - 4/30/30
URL: http://xulavoice.com